CLINICAL TRIAL: NCT06395779
Title: Comparison of Neuromuscular Exercises and Dance Therapy on Physical Performance and Kinesiophobia Results in Geriatrics
Acronym: NE-DTinGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ozum Cetinkaya, PT, MSC. ,Principal Investigator, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEDTGeriatrics
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Geriatrics; Neuromuscular Exercise; Dance Therapy; Kinesiophobia
Keywords: Geriatrics; Neuromuscular Exercise; Dance Therapy; Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Intervention Model Description: The study will be divided into two parallel groups: The neuromuscular exercise group and the Dance therapy group. Both groups will participate in exercise programs for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Exercise Group (Experimental): NE (Neuromuscular Exercise) group will participate in a 12-week exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns.
  Interventions: Behavioral: Neuromuscular Exercise Group
- Dance Therapy Group (Experimental): DT (Dance Therapy) Group will participate in 12-week dance training by a dance instructor. In dance therapy practices, simple and selected basic movements are appropriate to the level of the participants
  Interventions: Behavioral: Dance Therapy Group

INTERVENTIONS:
Behavioral: Neuromuscular Exercise Group — A 12-week Neuromuscular exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns will be created for the participants in Group 1.
  Arms: Neuromuscular Exercise Group
Behavioral: Dance Therapy Group — Participants in Group 2 will be given dance training by a dance instructor in the gym for 1 hour a day, 2 days a week, for a total of 12 weeks. In dance therapy practices, simple and basic movements are appropriate to the level of the participants, and special attention will be paid to the rhythm of the music not being fast. Latin dances were applied to the participants; selected rumba, merengue, bachata, and salsa movements. Dance therapy will start with a warm-up exercise (10 minutes), then dance exercises will be applied and the activity will end with a cool-down exercise (10 minutes).
  Arms: Dance Therapy Group

SUMMARY:
Objective: The aim of this study is to compare neuromuscular exercises and dance Therapy on physical performance and kinesiophobia results in geriatrics.

Methods: As a result of the power analysis (G-Power), 36 participants are planned to be included in this study Block randomization will be used to divide participants into 2 groups, each with at least 18 participants: Group 1 (NE Group) and Group 2 (DT Group) (Randomizer.org). NE (Neuromuscular Exercise) group will participate in a 12-week exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns.DT (Dance Therapy) Group will participate in 12-week dance training by a dance instructor. In dance therapy practices, simple and selected basic movements are appropriate to the level of the participants. Data will be collected using the Berg Balance Scale,30-second-Sit-to-Stand Test, Manual Muscle Testing, goniometer measurement and Tampa Scale of Kinesiophobia.

Practice Implications: This current study will contribute to the understanding of how neuromuscular exercises and dance therapy affect physical function and kinesiophobia in geriatrics.

DETAILED DESCRIPTION:
Human aging is a complex and individual process that occurs in biological, psychological, and social areas. The metabolic and physicochemical characteristics of cells gradually change with age, a process known as biological aging. This results in cellular self-regulation, regeneration, and structural alterations as well as the degeneration of healthy tissues and organs.

Physical performance impairments are linked to a wide range of negative health consequences, including osteoporosis, falls, and fractures, and are one of the most important health problems in geriatrics. Proprioceptive perception is significantly related to postural stability. Musculoskeletal system disorders (in physiological, neurological, kinesthetic, auditory, vestibular proprioception, and cognitive systems) cause balance problems, which may lead to an increase in the frequency of falls in the elderly.

Dance therapy is a physical and mental activity in which the body moves purposefully and rhythmically to music. Regardless of its type, dance brings physical, cognitive and spiritual goals. It includes physical goals such as effective and dynamic body mechanics, movement awareness and control, flexibility, strength, coordination, endurance and thus expanding the body's movement capacity.

Although the effects of dance therapy on strength, flexibility, stress, depression, quality of life, and sleep quality in geriatric patients have been investigated in the Turkish literature, no studies comparing dance therapy with any physical exercise program have been found. It is thought that this study will shed light on the literature in the mentioned field.

The aim of this study is to compare neuromuscular exercises and danceTherapy on physical performance and kinesiophobia results in geriatrics.

Methods:

Participants:

Volunteer individuals who met the inclusion and exclusion criteria and are first and second-year students of Alanya Alaaddin Keykubat University 60+ Renewal University will participate in the study. Detailed information about the study will be given to each participant who wishes to participate in the study, and their written and verbal consent will be obtained.

According to the power analysis made with the G-power program, it was found that 80% power can be obtained with 95% confidence when at least 30 people are included in the study. While calculating the sample size, timed get-up and walk test results [Group 1: 7.81 (standard deviation: 0.91), Group 2: 9.31 (standard deviation: 1.24)] were taken as a basis and the effect size was calculated as = 1.379. The risk of case loss was taken into account by taking a reserve rate of 20%, and it was planned to include 36 participants. The cases will be divided into 2 groups by block randomization using the internet program, consisting of at least 18 individuals: Group 1 [NE group] and Group 2 [AE group] (Randomizer.org).

Study Protocol:

The study will be divided into two parallel groups: The Neuromuscular Exercise group and the Dance Therapy group. Both groups will participate in exercise programs for 12 weeks.

Evaluations will be administered before and after exercise programs. Data will be collected using the Berg Balance Scale,30-second-Sit-to-Stand Test, Manual Muscle Testing, goniometer measurement, and Tampa Scale of Kinesiophobia.

Training and Exercise Applications:

A Neuromuscular exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns will be created for the participants in Group 1. Exercises will start with breathing and a 10-minute warm-up period, static and dynamic proprioception, kinesthesia training (weighting on the extremities, balance, walking, open kinetic chain, closed kinetic chain exercises), postural control exercises, Frenkel coordination exercises, balance exercises (balance ball). and with a balance board), muscle strength (calisthenic exercises, therabat exercises), plyometric exercises, and core stabilization exercises will be applied progressively over the weeks and will end with a 10-minute cooling period including flexibility and relaxation exercises.

2. Participants in Group 2 will be given dance training by a dance instructor in the gym for 1 hour a day, 2 days a week, for a total of 12 weeks. In dance therapy practices, simple and basic movements are appropriate to the level of the participants, and special attention will be paid to the rhythm of the music not being fast. Latin dances were applied to the participants; selected rumba, merengue, bachata, and salsa movements. Dance therapy will start with a warm-up exercise (10 minutes), then dance exercises will be applied and the activity will end with a cool-down exercise (10 minutes).

Exercise sessions in both groups will last 45-60 minutes and will be applied twice a week for 12 weeks. Blood pressure measurements of all participants will be taken before the applications. Exercise participation will be recorded in each session.

Statistical Analysis:

In the statistical analysis of data will obtain in this study, a Windows-based SPSS (IBM SPSS Statistics, Version 24.0, Armonk, NY, USA) package program will use. Continuous variables will express as a mean ± standard deviation or as a median (minimum-maximum values), and categorical variables as a number and percent. Analytical (Kolmogorov-Smirnov/Shapiro-Wilks test) and visual (Histogram and probability graphs) methods will use to test the conformity of data for normal distribution. When the parametric test assumptions were provided, Independent Sample T-Test will use to compare independent group differences; when the parametric test assumptions were not provided, the Mann Whitney-U test will use to compare independent group differences. In the dependent group analyses; when the parametric test assumptions were provided, Paired Sample T-Test will use; when the parametric test assumptions were not provided, Wilcoxon Test will use. Chi-Square Analysis and Fisher Exact Test will use compare differences between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Turkish,
* Being able to walk without using any assistive device,
* Being able to adapt to the training program and wanting to participate in the study voluntarily

Exclusion Criteria:

* Presence of neurological, musculoskeletal, inner ear or eye diseases that will cause functional disability and impaired standing balance,
* Those who have had changes in their medical treatments in the last 6 months,
* Those with a history of lower extremity surgery as it may affect balance tests,
* Volunteers who do not attend at least one of the training and evaluations for any reason.
* Volunteers who want to leave the study voluntarily.
* Volunteers who cannot continue working due to any additional disease that develops.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in balance | Before exercise programs and immediately after 12 weeks.
  Change in static balance will be evaluated using Berg Balance Scale. The scale consists of 14 questions scored between 0-4. Scores between 0-20 indicate imbalance, scores between 21-40 indicate normal balance, and scores between 41-56 indicate good balance.
Change in muscular fitness | Before exercise programs and immediately after 12 weeks.
  Change in muscular fitness will be evaluated using 30-second-Sit-to-Stand Test
Change in muscle strength | Before exercise programs and immediately after 12 weeks.
  Change in muscle strength will be evaluated using Manual Muscle Testing.
Change in range of motion | Before exercise programs and immediately after 12 weeks.
  Change in range of motion will be evaluated using Goniometer Measurement
Change in kinesiophobia | Before exercise programs and immediately after 12 weeks.
  Change in kinesiophobia will be evaluated using Tampa Scale of Kinesiophobia. The Scale consists of 17 questions and the high score indicates that the kinesiophobia is high.
Change in balance and walking | Before exercise programs and immediately after 12 weeks.
  Change in balance and walking will be evaluated using the Tinetti Balance and Gait Assessment. The first 9 of the 16 questions are about balance, and the next 7 questions are about walking. A score of 18 and below indicates a high risk of falling, a score of 19-24 indicates a moderate risk of falling, and a score of 24 and above indicates a low risk of falling.
Change of fear of falling | Before exercise programs and immediately after 12 weeks.
  Change in balance and risk of falling will be evaluated using alls Efficacy Scale International (FES-I). The Scale consists of 17 questions and the high score indicates that the fear of falling is high.

CONTACTS AND LOCATIONS:
Overall Officials: Özüm ÇETİNKAYA, PT, MSc, Principal Investigator — Alanya Alaaddin Keykubat University; Özgür NALBANT, Asst.Prof.Dr, Study Director — Alanya Alaaddin Keykubat University; Meriç ÖDEMİŞ, Dr., Study Chair — Alanya Alaaddin Keykubat University; Hatice GÜLSOY, Dr., Study Chair — Alanya Alaaddin Keykubat University
Locations (1):
- Özüm Çetinkaya, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva NC, Silva MC, Guimaraes MG, Nascimento MBO, Felicio LR. Effects of neuromuscular training and strengthening of trunk and lower limbs muscles in women with Patellofemoral Pain: A protocol of randomized controlled clinical trial, blinded. Trials. 2019 Oct 11;20(1):586. doi: 10.1186/s13063-019-3650-7. PMID 31604478
- [Background] Dziechciaz M, Filip R. Biological psychological and social determinants of old age: bio-psycho-social aspects of human aging. Ann Agric Environ Med. 2014;21(4):835-8. doi: 10.5604/12321966.1129943. PMID 25528930
- [Background] Esmail A, Vrinceanu T, Lussier M, Predovan D, Berryman N, Houle J, Karelis A, Grenier S, Minh Vu TT, Villalpando JM, Bherer L. Effects of Dance/Movement Training vs. Aerobic Exercise Training on cognition, physical fitness and quality of life in older adults: A randomized controlled trial. J Bodyw Mov Ther. 2020 Jan;24(1):212-220. doi: 10.1016/j.jbmt.2019.05.004. Epub 2019 May 7. PMID 31987547
- [Background] Sit RWS, Choi SYK, Wang B, Chan DCC, Zhang D, Yip BHK, Wong SYS. Neuromuscular exercise for chronic musculoskeletal pain in older people: a randomised controlled trial in primary care in Hong Kong. Br J Gen Pract. 2021 Feb 25;71(704):e226-e236. doi: 10.3399/bjgp20X714053. Print 2021. PMID 33495205
- [Background] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Derived] Cetinkaya O, Nalbant O, Odemis M, Gulsoy H. Effects of neuromuscular exercise and dance therapy on physical performance and kinesiophobia in GERIATRICS: A randomized controlled study. J Bodyw Mov Ther. 2025 Dec;45:545-554. doi: 10.1016/j.jbmt.2025.09.009. Epub 2025 Sep 19. PMID 41316619